CLINICAL TRIAL: NCT01147471
Title: Flail Chest: Early Operative Fixation Versus Non-operative Management - a Prospective Randomized Study
Brief Title: Flail Chest - Rib Fixation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: VCU-20100582
Record Dates: First submitted 2010-06-07; First posted 2010-06-22 (Estimated); Results first posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Flail Chest
Keywords: flail chest; rib fixation
MeSH Terms: conditions — Flail Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Operative rib fixation (Active Comparator): Randomized subjects will be operated upon within 72 hours of ventilation (early fixation) to stabilize the stove-in segment. Where all fractured ribs are accessible and the number of fractured ribs is few, stabilization of all fractured ribs would be the goal. However, where fractured ribs are in areas difficult to access, enough ribs, based on surgeon judgment, would be fixed to stabilize the stove-in segment. Post-operatively, the patients would receive the standard of care, similar to what is outlined for the non-operative arm.
  Operative fixation will be accomplished utilizing the MatrixRIB Fixation System (Synthes CMF, West Chester, PA, USA) according to the device's instructions for use. Sites will obtain the product based on their medical center's normal purchasing practices.
  Interventions: Device: operative rib fixation; Procedure: operative rib fixation surgery
- Non-operative arm (No Intervention): Randomized subjects to receive standard of care therapy for blunt thoracic trauma (as per each participating institution's own protocols):
  a. Ventilatory support b.Timing of extubation (removal from ventilator): c.Analgesia: institution should provide adequate analgesia utilizing available resources including oral, parenteral, epidural, local nerve blocks etc., d.Chest physical therapy, e.Postural drainage, f.Incentive spirometry - after extubation.

INTERVENTIONS:
Device: operative rib fixation — Randomized subjects will be operated upon within 72 hours of ventilation (early fixation)to stabilize the stove-in segment using a rib fixation system.
  Arms: Operative rib fixation
Procedure: operative rib fixation surgery
  Arms: Operative rib fixation

SUMMARY:
The purpose of this study is to determine whether operative fixation of unilateral flail chest provides greater benefit than non-operative treatment.

DETAILED DESCRIPTION:
Chest trauma is frequent in the multiply-injured patient and is directly responsible for 20-25% of trauma deaths. Additionally, chest trauma is a major contributory factor in another 25% of deaths after trauma. Besides short term mortality, injuries to the chest result in significant morbidity and cost of care and long term disability. Among patients sustaining chest trauma, flail chest is one of the more serious injuries. Patients require prolonged ventilation, ICU and hospital stays and have a high incidence of pulmonary infections. Survivors often go on to have significant impairment of pulmonary function and over half may never return to gainful employment.

The standard therapy of injuries to the chest wall, including flail chest has been effective analgesia, pulmonary toilet with postural drainage and aggressive chest physical therapy. Despite these measures, flail chest patients often do not do well. Early operative fixation (surgical anchoring and bracing of bones) to stabilize the chest wall and restore pulmonary dynamics has always been an attractive option. With improvements in patient selection, availability of good modern anesthesia and critical care, and mechanical fixation devices, small studies and several case reports testify to the feasibility of the concept and possible short and long term benefits. All but one small institutional study are retrospective in nature limiting the generalizability of the conclusions. In that small single institutional prospective trial in which patients with flail chest were randomized to either early operative fixation or standard non-operative therapy, patients randomized to early operative fixation showed significant improvements in both short- and long-term health outcomes resulting in lower in-hospital costs in the surgically treated group. Despite these very impressive results, although prospective, it is one study with a small number of patients from a single institution. The question of the benefits of operative fixation can only be conclusively answered by a larger multi-institutional prospective randomized study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults >21 years and <75 years
2. "Stove-in chest" to encompass both

   1. Unilateral flail chest (>3 ribs fractured at two places) or
   2. Contiguous rib fractures with at least 2 ribs pushed in > the rib diameter of the pushed in rib
3. Mechanically ventilated

Exclusion Criteria:

1. Patient unlikely to survive due to the trauma or age or multiple co-morbidities
2. Stove-in chest patients that do not require early (less than or equal to 48 hours of injury) ventilatory support
3. Bilateral flail chest
4. Sternal flail
5. P/F ratio < 200:1 over a period of greater than or equal to 6 hours while on the ventilator.
6. Other injuries that will likely prolong tracheal intubation and mechanical ventilation eg significant head injury resulting in low GCS (Glasgow Coma Score, a scale used to assess the central nervous system in patients who have undergone trauma), spinal cord injury resulting in paralysis of some or all of the respiratory muscles etc. These are merely examples. It is in the opinion of the investigator/surgeon what injuries would prolong tracheal intubation.
7. Any contra-indication to surgery including severe immunosuppression or severe chronic disease making elective surgery dangerous in the opinion of the surgeon
8. Inability to proceed with any aspect of critical care due to personal beliefs, living will etc eg non acceptance of blood products
9. Inability to obtain informed consent.
10. Subject's refusal for follow up
11. Pregnant women
12. Prisoners
13. Any other reason for which the potential subject is not a good candidate, in the opinion of the investigator.

If the site investigator believes that a patient is a good candidate for the study (i.e. requires ventilation primarily due to altered chest wall mechanics) but fails to meet all criteria, site may contact Dr Ajai Malhotra to see if a waiver will be granted.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajai K Malhotra, MD, Principal Investigator — Virginia Commonwealth University
Locations (7):
- United States (7):
  - Trauma Research & Education Foundation of Fresno, Fresno, California
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Board of Regents of the University of Oklahoma, Oklahoma City, Oklahoma
  - The University of Tennessee, Knoxville, Tennessee
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Nirula R, Allen B, Layman R, Falimirski ME, Somberg LB. Rib fracture stabilization in patients sustaining blunt chest injury. Am Surg. 2006 Apr;72(4):307-9. doi: 10.1177/000313480607200405. PMID 16676852
- [Background] Baker CC, Oppenheimer L, Stephens B, Lewis FR, Trunkey DD. Epidemiology of trauma deaths. Am J Surg. 1980 Jul;140(1):144-50. doi: 10.1016/0002-9610(80)90431-6. PMID 7396078
- [Background] Shorr RM, Mirvis SE, Indeck MC. Tension pneumopericardium in blunt chest trauma. J Trauma. 1987 Sep;27(9):1078-82. doi: 10.1097/00005373-198709000-00021. PMID 3656472
- [Background] LoCicero J 3rd, Mattox KL. Epidemiology of chest trauma. Surg Clin North Am. 1989 Feb;69(1):15-9. doi: 10.1016/s0039-6109(16)44730-4. PMID 2911786
- [Background] Shackford SR, Smith DE, Zarins CK, Rice CL, Virgilio RW. The management of flail chest. A comparison of ventilatory and nonventilatory treatment. Am J Surg. 1976 Dec;132(6):759-62. doi: 10.1016/0002-9610(76)90453-0. PMID 998864
- [Background] Relihan M, Litwin MS. Morbidity and mortality associated with flail chest injury: a review of 85 cases. J Trauma. 1973 Aug;13(8):663-71. doi: 10.1097/00005373-197308000-00001. No abstract available. PMID 4720987
- [Background] Landercasper J, Cogbill TH, Lindesmith LA. Long-term disability after flail chest injury. J Trauma. 1984 May;24(5):410-4. doi: 10.1097/00005373-198405000-00007. PMID 6716518
- [Background] Sankaran S, Wilson RF. Factors affecting prognosis in patients with flail chest. J Thorac Cardiovasc Surg. 1970 Sep;60(3):402-10. No abstract available. PMID 5271286
- [Background] Menard A, Testart J, Philippe JM, Grise P. Treatment of flail chest with Judet's struts. J Thorac Cardiovasc Surg. 1983 Aug;86(2):300-5. PMID 6876866
- [Background] Paris F, Tarazona V, Blasco E, Canto A, Casillas M, Pastor J, Paris M, Montero R. Surgical stabilization of traumatic flail chest. Thorax. 1975 Oct;30(5):521-7. doi: 10.1136/thx.30.5.521. PMID 1105874
- [Background] Thomas AN, Blaisdell FW, Lewis FR Jr, Schlobohm RM. Operative stabilization for flail chest after blunt trauma. J Thorac Cardiovasc Surg. 1978 Jun;75(6):793-801. No abstract available. PMID 661347
- [Background] Landreneau RJ, Hinson JM Jr, Hazelrigg SR, Johnson JA, Boley TM, Curtis JJ. Strut fixation of an extensive flail chest. Ann Thorac Surg. 1991 Mar;51(3):473-5. doi: 10.1016/0003-4975(91)90871-m. PMID 1998429
- [Background] Engel C, Krieg JC, Madey SM, Long WB, Bottlang M. Operative chest wall fixation with osteosynthesis plates. J Trauma. 2005 Jan;58(1):181-6. doi: 10.1097/01.ta.0000063612.25756.60. No abstract available. PMID 15674171
- [Background] Lardinois D, Krueger T, Dusmet M, Ghisletta N, Gugger M, Ris HB. Pulmonary function testing after operative stabilisation of the chest wall for flail chest. Eur J Cardiothorac Surg. 2001 Sep;20(3):496-501. doi: 10.1016/s1010-7940(01)00818-1. PMID 11509269
- [Background] Ahmed Z, Mohyuddin Z. Management of flail chest injury: internal fixation versus endotracheal intubation and ventilation. J Thorac Cardiovasc Surg. 1995 Dec;110(6):1676-80. doi: 10.1016/S0022-5223(95)70030-7. PMID 8523879
- [Background] Voggenreiter G, Neudeck F, Aufmkolk M, Obertacke U, Schmit-Neuerburg KP. Operative chest wall stabilization in flail chest--outcomes of patients with or without pulmonary contusion. J Am Coll Surg. 1998 Aug;187(2):130-8. doi: 10.1016/s1072-7515(98)00142-2. PMID 9704957
- [Background] Tanaka H, Yukioka T, Yamaguti Y, Shimizu S, Goto H, Matsuda H, Shimazaki S. Surgical stabilization of internal pneumatic stabilization? A prospective randomized study of management of severe flail chest patients. J Trauma. 2002 Apr;52(4):727-32; discussion 732. doi: 10.1097/00005373-200204000-00020. PMID 11956391
- [Background] Bastos R, Calhoon JH, Baisden CE. Flail chest and pulmonary contusion. Semin Thorac Cardiovasc Surg. 2008 Spring;20(1):39-45. doi: 10.1053/j.semtcvs.2008.01.004. PMID 18420125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients, 21 to 75 years old, admitted to the trauma unit with injuries that include either stove in chest (contiguous rib fractures with at least 2 ribs pushed in a distance greater than the rib diameter of the pushed in rib) or a unilateral flail chest (3 or more ribs fractures at two places). Patients must be on a ventilator.
Groups:
- Operative Rib Fixation: Randomized subjects will be operated upon within 72 hours of ventilation (early fixation) to stabilize the stove-in segment. Where all fractured ribs are accessible and the number of fractured ribs is few, stabilization of all fractured ribs would be the goal. However, where fractured ribs are in areas difficult to access, enough ribs, based on surgeon judgment, would be fixed to stabilize the stove-in segment. Post-operatively, the patients would receive the standard of care, similar to what is outlined for the non-operative arm.
  Operative fixation will be accomplished utilizing the MatrixRIB Fixation System (Synthes CMF, West Chester, PA, USA) according to the device's instructions for use. Sites will obtain the product based on their medical center's normal purchasing practices.
  operative rib fixation: Randomized subjects will be operated upon within 72 hours of ventilation (early fixation)to stabilize the stove-in segment using a rib fixation system.
Period: Through Initial Hospital Discharge
Arm/Group | Operative Rib Fixation | Non-operative Arm
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0
Period: Post-discharge Follow Up (Approx 2 Wks)
Arm/Group | Operative Rib Fixation | Non-operative Arm
Started | 13 | 11
Completed | 13 | 8
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — incarcerated | 0 | 1
Period: 3 Month Follow Up
Arm/Group | Operative Rib Fixation | Non-operative Arm
Started | 13 | 8
Completed | 12 | 6
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 1
Period: 6 Month Follow Up
Arm/Group | Operative Rib Fixation | Non-operative Arm
Started | 12 | 6
Completed | 8 | 4
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Population: Adult patients, 21 to 75 years old, admitted to the trauma unit with injuries that include either stove in chest (contiguous rib fractures with at least 2 ribs pushed in a distance greater than the rib diameter of the pushed in rib) or a unilateral flail chest (3 or more ribs fractures at two places). Patients must be on a ventilator.
Groups:
- Total: Total of all reporting groups
Arm/Group | Operative Rib Fixation | Non-operative Arm | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24
Mechanism of injury [Number; unit: participants]
  Fall from height | 1 | 0 | 1
  Motor cycle crash | 2 | 5 | 7
  Motor vehicle crash | 7 | 5 | 12
  Pedestrian struck | 3 | 1 | 4
Side & position of flail [Number; unit: participants]
  right side flail | 7 | 7 | 14
  left side flail | 6 | 4 | 10
  Postero-lateral | 10 | 9 | 19
  Antero-lateral | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Morbidity
Description: total days on ventilator, ICU length of stay, hospital length of stay
Time Frame: Measured daily during hospitalization (approx 1 month)
Population: analysis is the mean and standard deviation for # days spent on each item measured
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Operative Rib Fixation | Non-operative Arm
Number analyzed (Participants) | 13 | 11
days
  days on ventilator | 12.6 (8.5) | 7.0 (4.2)
  days in ICU | 23.1 (20.3) | 13.0 (6.1)
  days in hospital | 27.4 (18.7) | 20.8 (8.8)

2. Primary Outcome: Mortality
Description: Number of participants who died during any hospital stay.
Time Frame: Measured any time during hospital stay (approx 30 days)
Measure: Number; unit: participants
Arm/Group | Operative Rib Fixation | Non-operative Arm
Number analyzed (Participants) | 13 | 11
participants | 0 | 0

3. Secondary Outcome: Quality of Life
Description: Rand 36 health survey.
Time Frame: Measured at 3 and 6 months post-discharge
Population: Data not collected - insufficient participants completed follow up visits
Arm/Group | Operative Rib Fixation | Non-operative Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pulmonary Function
Description: Pulmonary function tests to measure forced vital capacity (FVC) and forced expiratory volume one (FEV1).
Time Frame: Measured at 3 and 6 months post-discharge
Population: Data not collected - insufficient participants completed follow up visits
Arm/Group | Operative Rib Fixation | Non-operative Arm
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Still on Narcotics at Post-discharge Follow-up
Description: Number of people still on narcotics at time of routine care post-discharge follow-up
Time Frame: approx 2 weeks post discharge
Measure: Number; unit: participants
Arm/Group | Operative Rib Fixation | Non-operative Arm
Number analyzed (Participants) | 12 | 8
participants | 7 | 6

ADVERSE EVENTS:
Time Frame: through 6 month post initial hospital discharge
Description: Only serious adverse events and related adverse events were collected.
Groups:
- Operative Rib Fixation: Randomized subjects will be operated upon within 72 hours of ventilation (early fixation) to stabilize stove-in segment. Where all fractured ribs are accessible and the number of fractured ribs is few, stabilization of all fractured ribs would be the goal. However, where fractured ribs are in areas difficult to access, enough ribs, based on surgeon judgment, would be fixed to stabilize stove-in segment. Post-operatively, the patients would receive standard of care, similar to what is outlined for the non-operative arm.
  Operative fixation will be accomplished utilizing the MatrixRIB Fixation System (Synthes CMF, West Chester, PA, USA) according to the device's instructions for use. Sites will obtain the product based on their medical center's normal purchasing practices.
  operative rib fixation: Randomized subjects will be operated upon within 72 hours of ventilation (early fixation)to stabilize the stove-in segment using a rib fixation system.
  operative rib fix
Arm/Group | Operative Rib Fixation | Non-operative Arm
Serious Adverse Events (participants affected / at risk) | 0/13 | 2/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operative Rib Fixation (N=13) | Non-operative Arm (N=11)
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — Unrelated.
cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) — unplanned hospitalization. Unrelated

LIMITATIONS AND CAVEATS:
Subject enrollment too low leading to insufficient data to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No